CLINICAL TRIAL: NCT03156205
Title: Effects of Patient-Directed Interactive Music Therapy on Sleep, Delirium and Melatonin Levels is Critically Ill Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2016-0873
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Critically Ill Adult Patients in Intensive Care Units
Keywords: critically ill patients; music therapy; sleep; delirium; melatonin; elderly
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interactive Music Therapy (Experimental)
  Interventions: Behavioral: interactive music therapy
- passive music listening (Other)
  Interventions: Behavioral: passive music listening
- passive earphone-use (Other)
  Interventions: Behavioral: passive earphone-use

INTERVENTIONS:
Behavioral: interactive music therapy — For the interactive music therapy intervention group, each patient received individual interactive music therapy sessions administered by professional music therapists during daytime; the patient participated in listening to music predetermined based on his/her preference during night time.
  Arms: Interactive Music Therapy
Behavioral: passive music listening — For the passive music listening group, each patient participated in music listening during night time without involving in interactive music therapy sessions during daytime.
  Arms: passive music listening
Behavioral: passive earphone-use — For the passive earphone use group (control group), each participant used headphone and eye mask without music listening at night time.
  Arms: passive earphone-use

SUMMARY:
(Background) Adults in intensive care units (ICU), especially elderly patients often suffer from a lack of sleep or frequent sleep disruptions due to physical, emotional stress such as pain, inflammation, and anxiety. Delirium, acute cognitive dysfunction, which result from sleep deprivation often leads to prolonged ICU stay and increase medical costs. Pharmacological and non-pharmacological interventions have been tried to improve the duration and quality of sleep and to maintain diurnal cycle. (Purpose) The aim of this study is to assess the efficacy of patient-driven interactive music intervention on sleep promotion in critically ill elderly adults. Delirium and urine/blood melatonin level will be assessed, too. In this study, randomized controlled trial for 50 elderly ICU patients who aged over 65 years in each group will be proceeded.

DETAILED DESCRIPTION:
Background: Adults in intensive care units (ICU), especially elderly patients often suffer from a lack of sleep or frequent sleep disruptions due to physical, emotional stress such as pain, inflammation, and anxiety. Delirium, acute cognitive dysfunction, which result from sleep deprivation often leads to prolonged ICU stay and increase medical costs. Pharmacological and non-pharmacological interventions have been tried to improve the duration and quality of sleep and to maintain diurnal cycle.

Purpose: The aim of this study is to assess the efficacy of patient-driven interactive music intervention on sleep promotion in critically ill elderly adults. Delirium and urine/blood melatonin level will be assessed, too. In this study, randomized controlled trial for 50 elderly ICU patients who aged over 65 years in each group will be proceeded.

Primary outcome: Richards-Campbell Sleep Questionnaire

Secondary outcome: Confusion Assessment Method - ICU, blood/urine melatonin level, ICU stay, Hospital stay, and mechanical ventilation duration / Delirium, acute cognitive dysfunction, which result from sleep deprivation often leads to prolonged ICU stay and increase medical costs. Elderly patients in ICU often suffer from a lack of sleep or frequent sleep disruptions due to physical, emotional stress such as pain, inflammation, and anxiety. Pharmacological and non-pharmacological interventions have been tried to improve the duration and quality of sleep and to maintain diurnal cycle. If interactive music therapy could improve quality of sleep and reduce incidence and severity of delirium in this patient population, it will be a good way to reduce medical costs without significant complications.

Expectation: There have been many trials to reduce delirium incidence and recover sleep patterns in ICU patients. If we could find interactive music therapy improve quality of sleep and reduce incidence and severity of delirium in this patient population, it will be a good way to reduce medical costs without significant complications. In addition, rhythm in music can be a appropriate support for respiration and motor function in elderly ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients aged over 65
* ASA(american society of anesthesiologists) class I-III

Exclusion Criteria:

* patients who had difficulties in communication
* history of neurological or psychiatric disorders, dementia, or alcohol use disorder.
* emergency surgery

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-09-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Richards-Campbell Sleep Questionnaire (RCSQ) | RCSQ will be measured for 3 days. (once/day)
  This scale evaluates sleep quality including perceptions of depth of sleep, sleep onset latency, number of awakenings, etc. It was designed as an outcome measure for assessment of the perception of sleep in critically ill patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim J, Choi D, Yeo MS, Yoo GE, Kim SJ, Na S. Effects of Patient-Directed Interactive Music Therapy on Sleep Quality in Postoperative Elderly Patients: A Randomized-Controlled Trial. Nat Sci Sleep. 2020 Oct 21;12:791-800. doi: 10.2147/NSS.S286375. eCollection 2020. PMID 33117015